CLINICAL TRIAL: NCT07292454
Title: Prevalence of Helicobacter Pylori on Patients With Chronic Inflammatory Bowel Disease (IBD) at the CHU of Guadeloupe
Acronym: HP-MICI
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Other Study IDs: PAP_RIPH2_2025/01
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: HELICOBACTER PYLORI INFECTIONS; Inflammatory Bowel Disease (Crohn's Disease and Ulcerative Colitis)
Keywords: intestinal microbioma; gastric microbioma; HELICOBACTER PYLORI INFECTIONS; Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Inflammatory Bowel Disease: Endoscopy is systematically performed in patients with Inflammatory Bowel Disease (IBD). In accordance with the recommendations of the French National Authority for Health, gastric biopsies are taken during digestive endoscopy as part of routine clinical care. Two additional biopsies (one fundic and one antral) are planned for research purposes, specifically for metagenomic analysis of the gastric microbiome.
  Interventions: Other: Biopsies

INTERVENTIONS:
Other: Biopsies — Gastric biopsies are taken during digestive endoscopy as part of routine clinical care. Two additional biopsies (one fundic and one antral) are planned for research purposes, specifically for metagenomic analysis of the gastric microbiome.

SUMMARY:
Clinical and experimental data suggest that dysbiosis may play a pivotal role in the pathogenesis of intestinal bowel disease (IBD). However, to the best of our knowledge, the composition of gastric and of intestinal microbiome has never been investigated in a population with IBD according to the presence/absence of Helicobacter pylori (H. pylori) in the stomach.

DETAILED DESCRIPTION:
H. pylori infection is one of the most widely spread infectious diseases in humans. Although the pathogenesis of IBD is unknown, this pathology could result from complex interactions between environmental factors and the intestinal microbiota, with dysbiosis likely being a key factor. In theory, H. pylori infection could be involved in the pathogenesis of IBD by inducing alterations in gastric and/or intestinal permeability or by causing immunological derangements. However, various studies indicate that the prevalence of H. pylori infection is low in patients with IBD, suggesting a protective role for this infection in the development of IBD.

The objective of the study is to investigate the potential link between H. pylori infection and IBD. Another objective is to analyze the complex interactions between the gastric and intestinal microbiome in a population with IBD according to the presence or absence of H. pylori in the stomach.

The study will be based on a prospective cohort of patients with IBD receiving medical care at the CHU of Guadeloupe.

ELIGIBILITY:
Inclusion Criteria:

Patients over 18 years old Patients with IBD from the CHU of Guadeloupe Patients benefiting from an investigation of H. pylori infection through gastric biopsies and/or serology at the time of diagnosis of IBD Patients affiliated to the French social security system Free informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research)

Exclusion Criteria:

Patients of less than18 years Patients having not given their writing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a confirmed diagnosis of Inflammatory Bowel Disease (Crohn's disease or ulcerative colitis) receiving routine follow-up care at the University Hospital of Guadeloupe. All participants are scheduled to undergo an upper gastrointestinal endoscopy as part of standard clinical management.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Prevalence of H. pylori infection in patients with Inflammatory Bowel Disease (IBD) | At the time of endoscopic evaluation (baseline only).
  Presence of Helicobacter pylori infection determined using gastric biopsies collected during clinically indicated upper gastrointestinal endoscopy. Infection status will be confirmed by standard histological assessment performed as part of routine care. The prevalence will be expressed as the proportion of IBD patients with confirmed H. pylori infection among all included IBD patients in the cohort.

SECONDARY OUTCOMES:
Demographic characteristics according to H. pylori infection status | Baseline.
  Comparison of demographic characteristics (age, sex, ethnicity) between IBD patients with and without confirmed H. pylori infection. Data collected at baseline from medical records.
Clinical characteristics according to H. pylori infection status | Baseline.
  Comparison of clinical characteristics (type of IBD, disease duration, clinical activity) between IBD patients with and without confirmed H. pylori infection. Data collected at baseline from medical records.
Biological inflammatory markers according to H. pylori infection status | Baseline.
  Comparison of biological markers related to disease activity (e.g., C-reactive protein, fecal calprotectin) between IBD patients with and without confirmed H. pylori infection.
IBD-related treatments according to H. pylori infection status | Baseline.
  Comparison of ongoing therapeutic regimens (e.g., immunosuppressants, biologics, corticosteroids) between IBD patients with and without confirmed H. pylori infection.
Prevalence of gastric intestinal metaplasia and dysplasia according to H. pylori infection status | Baseline.
  Histological assessment of gastric biopsies to determine intestinal metaplasia or dysplasia, compared between groups with/without H. pylori.
Composition of the gastric microbiome according to H. pylori infection status | Baseline.
  Metagenomic analysis of additional gastric biopsies (fundic + antral) to compare microbiome profiles between IBD patients with and without H. pylori.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de la Guadeloupe, Pointe-à-Pitre, CHU de La Guadeloupe, Guadeloupe

IPD SHARING:
Plan to Share IPD: Undecided